CLINICAL TRIAL: NCT00242528
Title: Open-label Study, to Evaluate the Safety and Tolerability of Zoledronic Acid in Patients With Bone Lesions Secondary to Multiple Myeloma.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EMX03
Record Dates: First submitted 2005-10-09; First posted 2005-10-20 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Myeloma
Keywords: Bone Lesions; Multiple Myeloma; zoledronic acid
MeSH Terms: conditions — Multiple Myeloma | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
To evaluate the safety and tolerability of intravenous zoledronic acid in the treatment of patients with multiple myeloma stage III with bone lesions related to Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
* Confirmed Diagnosis of Durie-Salmon Stage III Multiple Myeloma, with the following clinical characteristics:

A. At least 1 osteolytic bone lesion demonstrable in a conventional X-ray film. B. The patient will have to be receiving treatment for primary neoplasia, at the time of the start of this trial.

- Ambulatory patients aged ≥ 18 years.

Exclusion Criteria:

* Treatment with bisphosphonates in any moment during the last 12 months before visit 1. except for those patients that received only one dosis of bisphosphonates for any indication and when the administration has been 14 days before or older.
* Patients with an absence of a bone lesion clearly related to the primary cancer, and that is detectable in a conventional bone X-ray (simple film).
* Patients with a Serum Calcium level of ≤ 8 g/dl (2.00 mmol/L) or ≥ 12 mg/dL (3.00 mmol/L)
* Treatment with other investigational drugs within 30 days before inclusion in the trial.
* Serum Creatinine levels of > 3 mg/dl (265 umol/L).
* Total Billirubin levels of > 2.5 mg/dl (43 umol/L)
* Patients with a heart condition that has the NYHA criteria for a Grade III and IV functional class

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis